CLINICAL TRIAL: NCT01297179
Title: A Double-blind Two-sequence Crossover Study to Evaluate the Effect of Multiple Doses of YM178 on the Pharmacokinetics (PK) of an Ethinyl Estradiol and Levonorgestrel Containing Combined Oral Contraceptive (COC)
Brief Title: A Study to Evaluate the Possible Effects of Taking Mirabegron While Taking a Contraceptive Pill
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 178-CL-068; 2008-000216-32 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Volunteers; Pharmacokinetics of Mirabegron
Keywords: Pharmacokinetics; Oral contraceptives; Drug interactions; Pharmacokinetics of mirabegron
MeSH Terms: interventions — mirabegron; Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mirabegron — Oral
  Other Names: YM178
Drug: Minidril — Oral
  Other Names: ethinyl estradiol; levonorgestrel
Drug: Placebo — Oral

SUMMARY:
The objective of this study is to determine the effect of multiple doses of mirabegron on the pharmacokinetics of an oral contraceptive.

ELIGIBILITY:
Inclusion Criteria:

* Subjects above 35 years inclusive are re-evaluated for the risks of using of a COC
* Body Mass Index between 18.5 and 30.0 kg/m2, inclusive
* On oral contraceptive with 30ʯg ethinyl estradiol (EE) plus either 125ʯg or 150ʯg levonorgestrel (LNG) for at least three months prior to date of randomization and well tolerated
* During the study the subject is willing to use 1 of the 3 following contraceptive methods: diaphragm with spermicide, intrauterine device or partner is using condoms in combination with a spermicidal cream

Exclusion Criteria:

Subjects will be excluded from participation if any of the following apply:

* Known or suspected hypersensitivity to YM178 or any components of the formulation used
* Pregnant or breast feeding within 6 months before screening assessment
* Any of the liver function tests (i.e. ALT, AST and Alkaline phosphatase) above the upper limit of normal
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active Hay-fever)
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Abnormal pulse and/or blood pressure measurements at the pre-study visit as follows: Pulse <40 or >90 bpm; mean systolic blood pressure >140 mmHg; mean diastolic blood pressure >90 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically)
* A marked baseline prolongation of QT/QTc interval after repeated measurements of >450 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)
* Use of any prescribed or OTC (over-the-counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse within 3 months prior to admission to the Clinical Unit
* History of drinking more than 14 units of alcohol per week (1 unit = 270 cc of beer or 40 cc of spirits or 1 glass of wine) within 3 months prior to admission to the Clinical Unit
* Positive test for drugs of abuse or positive alcohol test on the day of admission into the clinical unit
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Clinical Unit
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2
* Subjects who, in the opinion of the investigator, are not likely to complete the trial for any reason
* Unwillingness to use additional barrier contraceptive methods for the course of the study and for one month after the end of study visit
* Any clinical condition, which, in the opinion of the investigator would not allow safe completion of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics of Ethinyl estradiol (EE) and Levonorgestrel (LNG) by analysis of blood samples. | Day 21 + Day 29

SECONDARY OUTCOMES:
Assessment of pharmacokinetics of mirabegron by analysis of blood samples. | Day 21 + Day 49

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Paris, France